CLINICAL TRIAL: NCT01820247
Title: Efficacy Study of Tripterygium Glycoside Combined With Enteral Nutrition in the Treatment of Crohn's Disease for Induction Remission
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhu Weiming (Other)
Responsible Party: Sponsor-Investigator, Zhu Weiming, vice director of General surgery institute, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD-IT1
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; enteral nutrition; Tripterygium Glycosides; induction remission
MeSH Terms: conditions — Crohn Disease | interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- enteral nutrition (Experimental): The patients receive treatment of enteral nutrition only.
  Interventions: Drug: enteral nutrition
- tripterygium glycosides (Experimental): The patients receive treatment of tripterygium glycosides only.
  Interventions: Drug: Tripterygium glycosides
- tripterygium glycosides and enteral nutrition (Experimental): The patients receive treatment of tripterygium glycosides and enteral nutrition.
  Interventions: Drug: enteral nutrition; Drug: Tripterygium glycosides

INTERVENTIONS:
Drug: enteral nutrition
  Arms: enteral nutrition; tripterygium glycosides and enteral nutrition
Drug: Tripterygium glycosides
  Arms: tripterygium glycosides; tripterygium glycosides and enteral nutrition

SUMMARY:
The purpose of this study is to assess the effect of Tripterygium Glycosides Combined with enteral nutrition in the treatment of Crohn's disease for induction remission and compare the therapeutic effect with patients who only received Tripterygium Glycosides or enteral nutrition.

DETAILED DESCRIPTION:
Crohn's disease is characterized by inflammation and ulceration of the small intestine and colon. Patients commonly experience abdominal pain, diarrhea，malnutrition and malaise which result in decreased quality of life and an increased risk of chronic disability and unemployment.

Tripterygium Glycosides(T2) is a chloroform/methanol extract Tripterygium wilfordii Hook F (TWHF), the traditional Chinese medicine,used in rheumatoid arthritis and nephritis. It has both immunomodulatory and anti-inflammatory activities.Our previous animal studies have revealed that the major component of T2, triptolide, could prevent the development of chronic colitis in interleukin-10 deficient mice. The phase I clinical trial in our institute also demonstrated that T2, or combined with enteral nutrition, is efficient for induction of remission in patients with active Crohn's disease.The common adverse effects of T2 are leucopenia,liver renal toxicity,oligospermia and amenorrhea.

The purpose of this study is to assess the effect of Tripterygium Glycosides Combined with enteral nutrition in the treatment of Crohn's disease for induction remission and compare the therapeutic effect with patients who only received Tripterygium Glycosides or enteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have a definitive diagnosis of Crohn's disease, based on WHO criteria
* Males and females ≥ 18 years old, including women who are not pregnant or lactating at the time of enrollment.
* Subjects should have a CDAI score ≥ 150 at week 0
* Able to swallow tablets
* Are capable of providing written informed consent and obtained at the time of enrollment
* Willing to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Bacterial,viral or other microbial infection(including HIV)
* Needing orally administered corticosteroids for the treatment of other diseases. Inhaled or dermatologic preparations are acceptable.
* Previous or current use of infliximab. current use of prescription doses or chronic/frequent use of NSAIDs
* Treatment with narcotic pain medications. (Anti-diarrheal agents such as loperamide and diphenoxylate are permitted)
* History of pancreatitis, except for subjects with a known but removed cause(such as gallstone pancreatitis)
* History of abnormal liver function tests, including AST or ALT >1.5 times upper limit of normal, alkaline phosphatase >2 times upper limit of normal, total bilirubin >2.5 mg/dL at screening (or within the previous 6 months, if known)
* History of malignancy
* Women who are pregnant or lactating at the time of enrollment, or who intend to be during the study period.
* Participation in other clinical trial within the past 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Therapeutic effect measured by CDAI and enteroscope | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- General Surgery Institute,Jinling Hospital,Nanjing,Jiangsu,China, Nanjing, Jiangsu, China